CLINICAL TRIAL: NCT03956082
Title: The Feasibility of Using the Ultravision™ System to Facilitate Low Impact Laparoscopic Surgery for the Treatment of Endometriosis
Brief Title: Ultravision™ System to Facilitate Low Impact Laparoscopic Surgery for Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, David Levine, Director Minimally Invasive Gynecology, Mercy Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-109
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Results first posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: This is a prospective single arm study. The study will enroll 20 patients. Comparisons to prior clinical trials and published literature will be made to assess the relative significance of the study results.
  Duration of Study: The target for the overall duration of the study is four months
Masking Description: A sample size of 20 patients should provide a sufficient sample size for comparative analysis to prior clinical data relative to Ultravision and published peer reviewed clinical data on laparoscopy and low impact laparoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- This is a prospective single arm study (Other): The Ultravision™ System is an FDA-cleared medical device that removes surgical smoke by means of electrostatic precipitation from the visual field during laparoscopic surgical procedures. "Surgical smoke" refers to the suspended particulate matter that is generated as a by-product of the combustion and other processes that are associated with the use of energy-based surgical instruments.
  Interventions: Device: Ultravision™ Visual Field Clearing System; Device: Ultravision Ionwand™

INTERVENTIONS:
Device: Ultravision™ Visual Field Clearing System — Laparoscopic surgery will be performed with the Ultravision Visual Field Clearing System. This system is indicated for the clearance of smoke and other particulate matter that is created during laparoscopic surgery. Ultravision Visual Clearing System removes surgical smoke by means of electrostatic precipitation
Device: Ultravision Ionwand™ — The Ionwand™ is introduced into the abdomen through either the Ultravision™ 5mm Trocar or a 2.5 mm percutaneous catheter. The Ionwand™ provides the source of electrons that create the negative ions that transiently charge the surgical smoke particles and accelerate their sedimentation.

SUMMARY:
This is a prospective single arm study. The study will enroll 20 patients. Comparisons to prior clinical trials and published literature will be made to assess the relative significance of the study results.The study will enroll patients indicated for laparoscopic surgery to treat endometriosis. Patients must meet all inclusion/exclusion criteria.

There are five main study objectives:

1. Demonstrate the feasibility of undertaking low impact laparoscopic surgery for endometriosis when using the Ultravision™ System.
2. Assess the impact of Ultravision on visual field clarity.
3. Determine the ability to complete the procedure while maintaining an abdominal pressure of < 10mmHg.
4. Quantify the consumption of CO2.
5. Collect data on additional clinical outcomes associated with the use of Ultravision and low impact surgery (i.e. end tidal CO2 levels (EtCO2), adverse events, cosmesis outcome, postoperative pain levels and pain medications).

DETAILED DESCRIPTION:
Background/Introduction: The Ultravision™ System is an FDA-cleared medical device that removes surgical smoke by means of electrostatic precipitation from the visual field during laparoscopic surgical procedures. "Surgical smoke" refers to the suspended particulate matter that is generated as a by-product of the combustion and other processes that are associated with the use of energy-based surgical instruments. Surgical smoke can obscure (partially or totally) the surgeon's view of the operative field and this has obvious safety implications for the patient. In the case of laparoscopic procedures, which are increasing in popularity, the smoke is retained within the "closed abdomen" and this, coupled with the CO2 pneumoperitoneum, presents additional challenges for the surgical team. The Ultravision™ System can therefore be considered an accessory to electrosurgical instruments to clear the surgical smoke generated during their use and as such will only be used when such devices are in use. The ability to operate at under "low impact" laparoscopic conditions has been shown by others to improve clinical outcomes by, for example, reducing post-surgical pain and with smaller incision sizes, improved cosmesis. For the purposes of this study "low impact" is defined as (1) a target pneumoperitoneal pressure of 10mm Hg; and (2) instead of 10mm and/or 12mm ports, the use of 3mm ports and one 5mm port. Using a standard insufflator, the combination of lower pneumoperitoneal pressure and smaller size ports creates visualization challenges for the surgeon due to the difficulty of preventing the buildup of surgical smoke within the abdomen. "Venting" or actively extracting the smoke through a trocar is known to be largely ineffective due to the narrow internal diameter of 3mm trocars, certainly unless the instrument is removed beforehand, which creates additional surgical challenges. Furthermore, operating under lower pressure can cause pneumoperitoneum to be lost upon venting of the smoke. The research question that is posed in this study is whether the Ultravision™ System, due to its unique mode of action which (unlike other smoke management approaches) provides smoke management without needing to extract or exchange CO2, provides effective visual field clearing, thereby facilitating low impact laparoscopic surgery when using a conventional insufflator. In addition, Ultravision™ does not require CO2 removal and replacement to achieve its intended use, thereby minimizing to the greatest extent possible patient CO2 exposure. CO2 is dry (effectively 0% relative humidity) and cold (typically 65F) and exposure is linked to postoperative pain and other adverse consequences such as patient cooling and tissue desiccation. Due its mode of action, Ultravision™ minimizes CO2 exposure to the patient. Laparoscopic surgery for the treatment of endometriosis is a common procedure for the removal of mild to moderate endometriosis. Diathermy is commonly used to remove the lesions which can be extensive, therefore this procedure presents an appropriate surgical procedure for this study. Assessments in terms of surgical field visualization, CO2 consumption, end tidal CO2, patient satisfaction for cosmesis, and postoperative pain will be conducted in order to determine if the Ultravision™ System is effective in enabling laparoscopic surgery under low impact laparoscopic conditions. Adverse event information will be reported. The study is an open label single arm study.

Study Purpose: There are five main study objectives:

1. Demonstrate the feasibility of undertaking low impact laparoscopic surgery for endometriosis when using the Ultravision™ System.
2. Assess the impact of Ultravision on visual field clarity.
3. Determine the ability to complete the procedure while maintaining an abdominal pressure of < 10mmHg.
4. Quantify the consumption of CO2.
5. Collect data on additional clinical outcomes associated with the use of Ultravision and low impact surgery (i.e. end tidal CO2 levels (EtCO2), adverse events, cosmesis outcome, postoperative pain levels and pain medications).

Study Hypothesis: The primary hypothesis being tested in this study is that Ultravision facilitates the utilization of low impact laparoscopic surgery techniques whilst maintaining an adequate visual field throughout the procedure with low demand for CO2 replenishment to maintain pneumoperitoneal pressure. Study Population The study will enroll patients indicated for laparoscopic surgery to treat endometriosis. Patients must meet all inclusion/exclusion criteria.

Study Design: This is a prospective single arm study. The study will enroll 20 patients. Comparisons to prior clinical trials and published literature will be made to assess the relative significance of the study results.

Study Endpoints: Success will be based on demonstration that the procedures using the Ultravision™ System achieves the following endpoints:

1. The ability to complete the procedure without increasing pneumoperitoneum due to visualization. Any increase beyond 10mm Hg and the reason for change will be recorded.
2. The quality of visualization in the laparoscopic field of view will be assessed by the investigator using a Visual Analog Scale (VAS).
3. Patient satisfaction in cosmesis outcome at the discharge follow-up visit assessed by means of a survey scaled from "very unsatisfied" to "very satisfied."
4. Patient postoperative pain assessments. Recorded by the patient each day from day 1 to day 7 postoperative using a 10 Numerical Rating Scale (NRS) where 0 is "no pain at all" to 10 "worst pain imaginable" and the location of the pain using a body diagram.
5. Amount and type of pain medication administered postoperatively. Recorded by the patient each day from day 1 to day 7 postoperative, and in person at final follow-up visit (study discharge visit).

Other Data Collection:

* End tidal CO2 volume (etCO2) (taken at the start of the procedure and at the completion of the procedure),
* Adverse Events,
* Electrosurgical instrument(s) used,
* Preoperative assessment: patient demographics, medical history, medication information, height and weight, pain (at intake visit)
* Estimate of case complexity/difficulty will be recorded. Study Size: A sample size of 20 patients should provide a sufficient sample size for comparative analysis to prior clinical data relative to Ultravision and published peer reviewed clinical data on laparoscopy and low impact laparoscopy.

Duration of Study: The target for the overall duration of the study is four months.

Data Analysis: Descriptive statistics for all endpoints will be applied to analyze the results.

Intended Use(per instructions for use): The Ultravision™ System is indicated for the clearance of smoke and other particulate matter that is created during laparoscopic surgery.

Device Description: The Ultravision™ System is an accessory to electrosurgical instruments that is used to clear the surgical smoke generated during their use and as such will only be used when such devices are in use. The system includes the following elements: Standalone battery-operated generator unit Ionwand™, which is introduced into the abdomen of the patient through either the Ultravision™ 5mm Trocar or a 2.5mm percutaneous catheter and provides the source of the electrons that create the negative ions that transiently charge the surgical smoke particles. Other accessories include a patient return adaptor and battery recharging station.

US Regulatory Status: The Ultravision™ System obtained regulatory clearance through US FDA's De Novo Classification Process (DEN 150022). The system has been in distribution in Europe since January 2014 and in the US since December of 2016, over 250 systems are currently in use. To date there have been no incident or medical device reports (patient injury reports) and there have been no product recalls.

Subject Identification & Selection: Potential subjects will be identified from the clinical practice of the participating investigator or by their respective research staff. Patients presenting to the clinical practice of the participating investigator for diagnosis or treatment consistent with the inclusion criteria will be informed about the study. With referral from the treating physician, patients scheduled for surgery prior to the start of the study may be contacted via telephone by a study team member to inform them of the study, assess their interest and assess their eligibility to participate. An IRB approved script will be used for such calls. For interested patients, a copy of the informed consent can be mailed or emailed to the patient for their review and consideration prior to their next clinic visit or the scheduled procedure. Each new subject presenting for evaluation or inclusion is to be assessed for adherence to the following inclusion/exclusion criteria. Determination of whether subjects satisfy the criteria may be established by review of medical records, subject interview, physical examination, or testing as appropriate. A baseline form is used to collect subject screening information and baseline assessments. Patients are considered enrolled once it has been demonstrated that the inclusion/exclusion criteria have been met and the patient signs the informed consent.

Subject Informed Consent: A partial waiver of HIPAA Authorization is being requested for the purposes of initial screening for study eligibility and recruitment purposes. Identifiable health information to be accessed under this waiver will include contact information, demographics, and medical history. Only study team members will have access to this information. Safeguards to maintain privacy and confidentiality of information will be taken as described in the data collection and management section of the protocol. Patient inclusion could be substantially hindered without the ability to review patients' records for eligibility and recruitment purposes, particularly for patients who may have already been scheduled for surgery at the time the study begins. Referred patients presenting for diagnosis or treatment consistent with the inclusion/exclusion criteria will undergo the informed consent process to authorize the gathering of data recorded on the Subject Screening & Enrollment Form. The study investigator will administer informed consent or may delegate the responsibility to a qualified individual as long as it is defined on the study responsibility log. When administering consent, it must be evident that the participant comprehends the nature of the study and the risks and benefits. Evidence is the patient is able to verbalize these topics in sufficient detail to confirm comprehension. Completion of the informed consent does not constitute enrollment. Enrollment occurs once screening is complete and all criteria for participation have been met. Subjects must document their consent for study participation by signing the Institutional Review Board approved Informed Consent Form. The informed consent process must be consistent with the Declaration of Helsinki. The subject must be given the opportunity to ask questions of, and receive answers from, study personnel prior to a request to sign the Informed Consent Form. This form is to be co-signed by the investigator. Failure to obtain consent prior to subject participation is considered a protocol deviation and must be reported to the Institutional Review Board. After the subject and investigator sign the Informed Consent Form, the original is to be filed in the subject's study binder. Copies will be filed in the subject's medical record and the subject is also to be given a copy.

Screening & Enrollment: Patient demographics and other baseline information will be collected to establish whether the patient meets the requirements for the study. It is assumed that a physical exam will be conducted as part of the standard of care. Each patient will be assigned a unique study number. Baseline information will be collected, consistent with the standard of care. Baseline assessment is conducted at the preoperative visit.

Procedure Protocol: The device is used in accordance with the instructions for use. An initial target pneumoperitoneal pressure setting of 10mmHg will be used for the procedure. At the discretion of the surgeon investigator, pressure will be adjusted as needed to accomplish the surgical procedure. A standard insufflator with 3mm ports and one 5 mm ports will be used for the procedure.

Surgeon Survey: Immediately post procedure the investigator will be asked to provide feedback regarding visibility, smoke management and complexity of the procedure.

1. Overall quality of visualization (responses will be recorded on a VAS scale).
2. How often was smoke management a negative factor during the procedure (responses will be recorded on a VAS Scale).
3. Complexity of the procedure (simple, routine or complex).

Post Procedure Follow-Up Protocol: Post-operative days 1-7:

Subjects will be asked to complete a daily diary/self-assessment of pain. Assessment will include a pain rating, location of pain and medications taken for pain. The diary/self-assessment is included as a separate document.

Post-operative 2 week (± 3 days) follow up visit: A 2 week follow up visit is current standard of care. At this visit, adverse events will be assessed. A final pain assessment will be administered during this visit.

Post-operative 4 week (± 1 week) follow up phone call: Patient satisfaction for cosmesis (scar appearance) after the surgery will be collected by means of a telephone follow-up where a simple cosmesis satisfaction survey will be administered by a study team member.

Adverse Event Categories: For purposes of this protocol the adverse event definitions are derived from Good Clinical Practice (GCP) standards and FDA Guidance. The signs, symptoms, and sequelae of an underlying adverse event (linked pathophysiologically to the AE) should not be reported as separate adverse events. All adverse events, of any type, are to be recorded on an "Adverse Event Form". Adverse events are to be characterized by their severity, relatedness the implant procedure, need for therapy, and resolution status. Adverse events will initially be characterized as "serious" or "non-serious" by the study investigator.

Adverse Event Adjudication: Events are to be initially judged by the investigator as to their relatedness to the study device, surgical procedure, or "other etiology". The classifications will be "not related", "probably not related", "undetermined", "probably related", or "related".

Reporting of Adverse Events and Unanticipated Problems: Serious adverse events and Unanticipated Problems related to the research will be reported to the Mercy Institutional Review Board.

Subsequent Surgical Interventions: Some complications may lead to a subsequent surgical intervention. The reason for each subsequent surgical intervention and the action taken is recorded on the case report form, along with the identification of the type subsequent surgical interventions according. The exact type of intervention must be specified.

Patient Withdrawal: A patient may choose to withdraw from participation in the study at any time without penalty. If a patient chooses to withdraw, they will still receive medical care consistent with the standard of care. The investigator may at their discretion withdraw a patient from participation or where intraoperative exclusions (defined in the I/E criteria) occur. Other examples include if the procedure necessitates conversion from laparoscopic to open technique, lack of adherence to visit schedule, adverse events, or safety concerns. For all withdrawals the date, point in the study, and reason for withdrawal will be recorded. Patients that withdraw prior to the procedure or are withdrawn from the study due to an intraoperative exclusion are replaced.

Study Suspension/Termination: If for any reason the principle investigator chooses to suspend or terminate the study, the IRB shall be informed of the decision and the basis of the decision.

Provision and Inventory of Study Devices: The device and required materials will be provided to the Investigator by Alesi Surgical Ltd.

Data Collection and Management: The investigator and study team members as delegated are responsible for collecting the data from the study.

Imaging Diagnostics: All imaging performed for patients is considered consistent with standard of care.

Sample Size Justification: Ultravision is already cleared by the FDA for use in laparoscopic endometriosis. This post-market study is intended to evaluate user satisfaction and the relative impact the Ultravision™ System has on the procedure as opposed to demonstrating safety and efficacy. The sample size selected (20) is considered to be a sufficient quantity to establish whether or not low impact surgery is facilitated with the use of the Ultravision™ System. This is designed as a single arm study to demonstrate feasibility of device use under low impact laparoscopy. The Ultravision will either enable the procedure to be completed as planned or not, therefore a control arm is not considered necessary to make this determination. In addition, incorporating a control arm using the same conditions without the use of Ultravision may not be in the best interest of the patient. The study design is considered to appropriate for the research question that is being posed.

Data Analysis: Data collected will be summarized using descriptive statistics. Results from other studies conducted by Alesi as well as clinical data gleaned from the medical literature will be used to assess the relative significance of the study results. Additional exploratory analysis may be conducted during data analysis.

Training Procedures: The Principal Investigator in the study is a current Ultravision user, no additional device training is required. To ensure compliance with the study plan and regulatory requirements as well as accurate data collection, site training will include a detailed review of this Investigational Plan, case report form (CRF) completion instructions, adverse event reporting, device handling and inventory, monitoring logistics, and regulatory requirements.

Administration: This study is being conducted as an "Investigator Sponsored" post-market study. The Investigator holds ultimate responsibility for the design, conduct, analysis, and reporting of the results from this study and is the primary contact for all matters related to this investigational plan. The Primary Investigator is also accountable for monitoring this investigation and performing those actions necessary to protect the scientific credibility of the way this study is conducted.

Regulatory Compliance: The Principal Investigator is responsible for ensuring that the study is implemented at their site according to the Investigator Agreement, this protocol, applicable laws, regulations, and any conditions of approval by either the respective Institutional Review Board. The Principal Investigator is also responsible for ensuring that this study is conducted in a scientifically credible and ethical manner. The Principal Investigator is responsible for the selection, training, and supervision of site-specific research personnel. The Principal Investigator shall always perform responsibilities in a manner which protects the rights, safety, and well-being of subjects. The Principal Investigator and all research staff participating in this investigation are expected to adhere to this investigational plan, Good Clinical Practices, applicable privacy laws, the Declaration of Helsinki, and any approval requirements imposed by an Institutional Review Board. The study will be submitted for review and approval by the Mercy Institutional Review Board.

Privacy and Confidentiality: This study is to be performed in accordance with all applicable privacy laws. All data and information concerning subjects and their participation in this trial are considered confidential. Only authorized investigators and approved study personnel will have access to some portions of these confidential files. Institutional Review Boards and other regulatory authorities also have the right to inspect and copy records pertinent to this trial.

Investigator Records: Records to be maintained by the investigator in a designated study file include: Site information: Site signature log, Responsibility log, Training and credentials of study personnel.

Device information: Ultravision and diathermy device inventory log including: date, quantity, lot numbers of all devices, identification of all persons the device was used on, and final disposition, Shipping documents.

Clinical study Plan/Protocol: Plan and all amendments. Institutional Review Boards Records: Institutional Review Board Membership List, Submission to Institutional Review Boards, Approval letters, Notification of unanticipated adverse device events, updates/reports, Any other communication.

Screening and enrollment form, Consent Form: Institutional Review Boards approved copy, Revised approved, consent forms.

Case Report Forms (CRFs): Annotated CRF and/or CRF instructions (if applicable), Blank CRFs and completion instructions (if applicable) Correspondence: All correspondence of material concern relating to the trial between the investigator and other parties (e.g. IRB).

The following records must be maintained for each subject enrolled in the trial:

Signed Consent Form, Completed CRFs, Protocol Deviation Forms, Complete medical records, including procedure reports, lab reports, professional notes, etc. for participating subjects. Records pertaining to subject death during the investigation (including death records, death certificate, and autopsy report, if performed).

Risk/Benefit Assessment: Medical treatment provided to the patient is within the standard of care for this type of procedure. Additional assessments for procedure data, end tidal CO2 measures, post procedure pain assessments, pain medication, cosmesis result, and adverse event information do not introduce new risks to the patient. If necessary, the investigator will increase the pressure required to achieve adequate visualization/working space.

As surgical accessory devices, the Ultravision does not administer any medical treatment. The risks associated with its use are consistent with other surgical accessories used in laparoscopic surgery. The Ultravision™ System is required to undergo testing for sterility, biocompatibility, and electrical safety in order to demonstrate that such risks have been mitigated to acceptable levels. The benefits that are being evaluated in this study are quality of visualization under low impact laparoscopic conditions with the anticipated improvement in patient outcomes in terms of cosmesis and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST meet all the following:

Is 18 years or older.

* Provide written informed consent prior to trial procedures after studies indicate that the patient needs the prescribed procedure.
* Agrees to attend all follow-up assessments.
* Is indicated for laparoscopic surgery for the treatment of endometriosis.
* Able to read and understand English.

Exclusion Criteria:

Subjects MUST not have any of the following:

* Existing comorbidities that would contraindicate them for laparoscopic surgery.
* Patient anatomy that is not compatible with the use of the Ionwand catheter i.e. abdominal wall thickness that exceeds the working length of the Ionwand catheter identified intraoperatively
* Patient with a BMI > 50
* Be pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will enroll female patients who are indicated for laparoscopic surgery for the treatment of endometriosis
Enrollment: 15 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Minimally Invasive Gynecology, Mercy Hospital St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- This is a Prospective Single Arm Study: The Ultravision™ System is an FDA-cleared medical device that removes surgical smoke by means of electrostatic precipitation from the visual field during laparoscopic surgical procedures. "Surgical smoke" refers to the suspended particulate matter that is generated as a by-product of the combustion and other processes that are associated with the use of energy-based surgical instruments.
  Ultravision System: Laparoscopic surgery will be performed with the Ultravision Visual Field Clearing System. This system is indicated for the clearance of smoke and other particulate matter that is created during laparoscopic surgery. Ultravision Visual Clearing System removes surgical smoke by means of electrostatic precipitation
Period: Overall Study
Arm/Group | This is a Prospective Single Arm Study
Started | 15
Completed | 9
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 9
Age, Customized [Median (Full Range); unit: years]
  Age of participants | 28 [20 to 48]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Women | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9
Body Mass Index (BMI) [Median (Standard Deviation); unit: kg/m^2] | 24.5 (4.7)
Endometriosis diagnoses [Count of Participants; unit: Participants]
  Pelvic pain | 4
  Ovarian cyst | 2
  Other (diagnoses included menorrhagia, hematochezia and dysmenorrhea and dyspareunia) | 3
Indicated pain location on representative human figure [Count of Participants; unit: Participants]
  Not applicable | 5
  Lower abdomen | 2
  Left lower quadrant (LLQ) | 1
  Right lower quadrant (RLQ) | 1
Pain score on a scale from 0 (no pain) to 10 (worst pain imaginable). [Count of Participants; unit: Participants]
  Pain score of 0 | 5
  Pain score of 1 | 2
  Pain score of 2 | 1
  Pain score of 3 | 1
Recorded name, dose and frequency of any pain medication taken within 24 hours of surgical procedure [Count of Participants; unit: Participants]
  Taking "1/2 pill" Percocet (class 4 drug) (not prescribed) prn for pain within 24 of surgery. | 1
  Taking 600mg ibuprofen (class 2 drug) prn for pain within 24 of surgery. | 1
  Not taking pain medication within 24 hours of surgery. | 5
  Unspecified pain medication for unrelated condition(s) | 2

OUTCOME MEASURES:

1. Primary Outcome: Procedure Completed Without Change in Intra-abdominal Pressure
Description: The ability to complete the procedure without increasing pneumoperitoneum due to visualization. Any increase beyond 10mm Hg and the reason for change will be recorded.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Quality of Visualization Laparoscopic Field
Description: The quality of visualization in the laparoscopic field of view will be assessed by the investigator using a Visual Analog Scale (VAS). The scale will rate the overall quality of visualization during the procedure on a scale numbered 0 to 100, in increments of 10, where 0 equals poor and 100 equals excellent.
Time Frame: Intra-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 9
score on a scale | 100 (0)

3. Secondary Outcome: Cosmesis Outcome
Description: Patient satisfaction in post-surgical cosmesis outcome, administered via telephone, assessed by means of a survey scaled from 1 - 7, where 1 = "very unsatisfied" and 7 = "very satisfied".
Time Frame: A mean of 31 days (SD=2.8) after surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 9
Participants
  5 | 1
  6 | 2
  7 | 6

4. Secondary Outcome: Postoperative Shoulder Pain Assessment (Day 1-7)
Description: Patient shoulder postoperative pain assessments. Recorded by the patient each day from day 1 to day 7 postoperative using a 10 Numerical Rating Scale (NRS) where 0 is "no pain at all" to 10 "worst pain imaginable".
Time Frame: Day 1-7 postoperative
Population: The pain diary for post-operative days 1-7 was completed by eight of the nine subjects.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 8
score on a scale
  Post-operative day 1 | 3.125 [0 to 7]
  Post-operative day 2 | 1.25 [0 to 5]
  Post-operative day 3 | 0.5 [0 to 2]
  Post-operative day 4 | 0.625 [0 to 3]
  Post-operative day 5 | 0.25 [0 to 2]
  Post-operative day 6. | 0.125 [0 to 1]
  Post-operative day 7 | 0 [0 to 0]

5. Secondary Outcome: Opioid/Opioid-containing Medication Taken Postoperatively for Pain
Description: Some subjects recorded taking opioid and non-opioid medications for pain. Non-opioid medications included non-steroidal anti-inflammatory drugs and acetaminophen.
Time Frame: Day 1-7 postoperative
Population: The pain diary for post-operative days 1-7 was completed by eight of the nine subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 8
Participants
  Post-operative day 1 | 5
  Post-operative day 2 | 3
  Post-operative day 3 | 0
  Post-operative day 4 | 0
  Post-operative day 5 | 0
  Post-operative day 6 | 0
  Post-operative day 7 | 1

6. Other Pre Specified Outcome: End Tidal CO2 Volume
Description: End tidal CO2 volume (etCO2) taken at the start of the procedure and at the end of the procedure (trocar removal).
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 9
mm Hg
  At the beginning of the procedure. | 32.1 (3.1)
  At the end of the procedure. | 35.2 (2.4)

7. Other Pre Specified Outcome: Case Complexity
Description: Estimate of case complexity/difficulty will be recorded using a Visual Analog Scale (VAS) indicating how often smoke management was a factor during the procedure on a scale ranging from 1 - 100, where 1 was "Often" and 100 was "Never".
Time Frame: End of procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 9
score on a scale | 100 (0)

8. Secondary Outcome: Postoperative Abdominal Pain Assessment (Day 1-7)
Description: Patient postoperative abdominal pain assessments. Recorded by the patient each day from day 1 to day 7 postoperative using a 10 Numerical Rating Scale (NRS) where 0 is "no pain at all" to 10 "worst pain imaginable".
Time Frame: Day 1-7 postoperative
Population: The pain diary for post-operative days 1-7 was completed by eight of the nine subjects.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 8
score on a scale
  Post-operative day 1 | 3.125 [0 to 6]
  Post-operative day 2 | 3.75 [1 to 6]
  Post-operative day 3 | 3 [1 to 5]
  Post-operative day 4 | 2.75 [1 to 6]
  Post-operative day 5 | 2.25 [1 to 4]
  Post-operative day 6 | 1.6875 [0 to 7.5]
  Post-operative day 7 | 1.375 [0 to 3]

9. Secondary Outcome: Non-opioid Medication Taken Postoperatively for Pain
Description: as for outcome 5
Time Frame: Day 1-7 postoperative
Population: The pain diary for post-operative days 1-7 was completed by eight of the nine subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | This is a Prospective Single Arm Study
Number analyzed (Participants) | 8
Participants
  Post-operative day 1 | 6
  Post-operative day 2 | 7
  Post-operative day 3 | 5
  Post-operative day 4 | 6
  Post-operative day 5 | 4
  Post-operative day 6 | 3
  Post-operative day 7 | 3

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | This is a Prospective Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | This is a Prospective Single Arm Study (N=9)
Shoulder pain (Injury, poisoning and procedural complications) | 5 (14)
Abdominal pain (Injury, poisoning and procedural complications) | 9 (60)
Pain at unspecified location (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT03956082/Prot_001.pdf